CLINICAL TRIAL: NCT01124422
Title: A Study of Fluticasone Propionate/Salmeterol DISKUS Combination Product 250/50 mcg Twice Daily Plus Tiotropium 18 mcg Daily Versus Placebo DISKUS Twice Daily Plus Tiotropium 18 mcg Daily on Exercise Time and Physiological Parameters in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Fluticasone Propionate/Salmeterol Combination 250/50 DISKUS in the Exercise Endurance Time in Patients With Chronic Obstructive Pulmonary Disease
Acronym: ESWT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113877
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: endurance shuttle walk test; chronic obstructive pulmonary disease; fluticasone propionate; dyspnea; exercise endurance time; tiotropium; salmeterol; exercise inspiratory capacity; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone propionate/salmeterol DISKUS 250/50 + tiotropium (Experimental): This is the active DISKUS (that is, containing fluticasone propionate/salmeterol combination) + open-label tiotropium
  Interventions: Drug: fluticasone propionate/salmeterol inhalation powder DISKUS 250/50; Drug: tiotropium bromide inhalation powder HandiHaler
- placebo DISKUS + tiotropium (Placebo Comparator): This is the DISKUS and excipient minus the active ingredient (which is fluticasone propionate/salmeterol combination) + open-label tiotropium
  Interventions: Drug: tiotropium bromide inhalation powder HandiHaler

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol inhalation powder DISKUS 250/50 — Experimental comparator consisting of inhaled corticosteroid plus long-acting beta agonist combination also known as ADVAIR DISKUS
  Arms: fluticasone propionate/salmeterol DISKUS 250/50 + tiotropium
Drug: tiotropium bromide inhalation powder HandiHaler — Open-label drug also known as Spiriva HandiHaler

SUMMARY:
The objective of this study is to demonstrate that, when added to tiotropium (TIO), fluticasone propionate/salmeterol combination (FSC) DISKUS 250/50 significantly increases exercise endurance time (EET) in the endurance shuttle walk test (ESWT), compared to TIO alone. Male and female subjects at least 40 years of age with a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) are eligible. Subjects will be screened and consented at or during a 6-week (wk) period prior to visit (V)1. The 4-wk run-in period begins immediately after V1, when subjects receive open-label TIO plus as-needed relief inhaler (identical formulations called albuterol in the US and salbutamol in Canada). At V2, subjects will perform an incremental shuttle walk test (ISWT) to establish their maximal walk response. The first ESWT will occur at V3. Subjects must demonstrate an EET of ≤20 min that is reproducible (EET from V3 and V4 varying by ≤2 min). Eligible subjects are then randomized at V5 to either FSC 250/50mcg DISKUS twice daily plus open label TIO 18 mcg daily, or placebo DISKUS twice daily plus open label TIO 18 mcg daily for the 4-wk treatment period. The last study visit is V6. The primary efficacy measure is the difference between the EET at V6 (wk-8) vs. V4 (wk-3; the last ESWT done before randomized study drug is given). Secondary efficacy measures include V6 vs. V4 comparisons in exercise dyspnea scale (EDS), exercise inspiratory capacity (EIC) and cardio-respiratory measurements (CRM), and V6 vs. V5 comparisons in dyspnea related to activities of daily living (baseline dyspnea index and transition dyspnea index interviewer-administered [BDI-TDI]) and quality of life (Chronic Respiratory Disease Questionnaire Self-administered Standardized [CRQ-SAS]). The safety measure will be an assessment of adverse events. We will also attempt to validate prospectively the minimal clinically-important difference (MCID) for a change in the EET through correlation with dyspnea and quality of life results.

DETAILED DESCRIPTION:
We postulate that adding fluticasone propionate/salmeterol combination DISKUS 250/50 (FSC) to tiotropium (TIO) will improve exercise endurance time (EET) and its clinical and physiologic correlates, based on the combination of the three different mechanisms of action represented. We propose to test this hypothesis by comparing outcomes of exercise testing (Endurance Shuttle Walk Test; ESWT) with FSC added to TIO compared to those on TIO alone.

The primary objective is to demonstrate that, when added to TIO, FSC significantly increases EET compared to TIO alone at Visit 6 (V6; week [wk]-8) vs. V4 (wk-3; the last ESWT before double-blind drug).

Secondary efficacy measures will be as follows. Exercise dyspnea scale (EDS), exercise inspiratory capacity (EIC) and cardio-respiratory measurements (CRM) will involve V6 vs. V4 comparisons. Dyspnea related to activities of daily living (ADLs) will be assessed using the baseline dyspnea index and transition dyspnea index interviewer-administered (BDI-TDI), and quality of life will be assessed using the Chronic Respiratory Disease Questionnaire Self-Administered Standardized (CRQ-SAS). The BDI-TDI and CRQ-SAS will be based on comparisons of data from V6 vs. V5. We will also attempt to validate prospectively the minimal clinically-important difference (MCID) for a change in the EET through correlation with dyspnea (Likert scale).

Safety evaluations will include the type, incidence and severity of adverse events.

This is a randomized, parallel-group study totalling 6 visits. Screening is at or up to 6 wk prior to V1, and includes a discussion of study procedures, a review of inclusion/exclusion criteria, collection of informed written consent, adjustment of medications and determination of spirometry pre- and post-albuterol/salbutamol. At V1, subjects meeting inclusion criteria will be enrolled, familiarized with the incremental shuttle walk test (ISWT), and given paper diaries.

The run-in will begin with the dispensing of open-label medications at the end of V1. During the 4-wk run-in, subjects will have 3 visits (V2-V4). Open-label TIO will be taken daily beginning after V1, and open-label relief inhaler (identical formulations called albuterol in the US and salbutamol in Canada) will be taken on an as-needed basis beginning after V1. Open-label medications will be withheld before V2, V3 and V4 (last dose of TIO, the morning of the day before the visit; last dose of albuterol/salbutamol, at least 6 hr before the start of the visit). At V2, subjects will be given open-label TIO, will undergo ISWT 2.5-hr post-TIO, and will be familiarized with the ESWT. At V3 and V4, subjects will be given open-label TIO, and will undergo ESWT 2.5-hr post-TIO. ESWT will be performed again at V4 only if the EET at V3 was ≤20 min. Subjects will be studied at V5 if the EET result from V4 is also ≤20 min and the EET from V3 and V4 vary from each other by ≤2 min; otherwise, subjects will be withdrawn. The ESWT from V4 will be used as the baseline EET for exercise-related outcomes because it will be the last ESWT done before double-blind study drug is given.

Open-label medications will be withheld before V5 and V6 (last dose of TIO the morning of the day before the visit; last dose of albuterol/salbutamol, at least 6 hr before the start of the visit). At V5, subjects will undergo spirometry, lung volumes and diffusing capacity, and will be randomized. Subjects will then be given open-label TIO and double-blind DISKUS study drug, and undergo spirometry and lung volumes 2 hr post-TIO/double-blind DISKUS study drug, and ESWT 2.5 hr post-dose. Per randomization, subjects will receive for 4 wk after V5, open-label TIO plus either FSC or placebo DISKUS. Double-blind DISKUS study drug will be withheld before V6 (last dose the evening of the day before the visit). V6 will be the last study visit, consisting of spirometry and lung volumes, followed by open-label TIO and double-blind DISKUS study drug, spirometry and lung volumes 2 hr post-dose, and the final ESWT 2.5 hr post-dose.

All study visits will begin with a check-up to determine eligibility for further study procedures. Details of the paper diary report will be reviewed after drug administration, V2 through V6. Immediately after review of the paper diary, BDI (at V5), TDI (at V6) and CRQ-SAS (V5 and V6) will be undertaken, and the post-dose study activities, as outlined above, will follow.

Final contact will be by telephone approximately 2 wk after V6 or Early Withdrawal. The total duration of the study will be 8 wk, including the 4 wk run-in and the 4 wk period of double-blind plus open-label treatment. There will also be a screening period of up to 6 wk prior to V1, and the 2-wk period after the final study visit for phone call follow-up.

Subjects at a subset of sites will undergo EIC and CRM during each ESWT using portable telemetric monitoring (Oxycon Mobile; CareFusion, San Diego, CA).

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria at V1.

* Consent: A signed and dated written informed consent must be obtained from the subject and/or subject's legally acceptable representative prior to study participation.
* Age: at least 40 yr of age
* Sex: Male or Female

Females are eligible to participate only if they are currently not pregnant and not lactating. In addition, female subjects should not be enrolled if they plan to become pregnant during the time of study participation. A female is otherwise eligible to enter and participate in the study if she is of:

* non-child bearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal); or,
* child-bearing potential, has a negative pregnancy test (urine) at screening, and is committed to the consistent and correct use of an acceptable method of birth control, starting at V2, throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of six days), as defined by at least one of the following:
* use of implants of levonorgestrel or etonogestrel
* percutaneous contraceptive patches
* use of injectable progestogen
* use of oral contraceptive (either combined estrogen/progestin or progestin only)
* use of any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per yr
* male partner is sterile (vasectomy with documentation of azoospermia; note that a verbal report of azoospermia is acceptable) and is the sole sexual partner for that female subject prior to the female subject's entry into the study
* double-barrier method; condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicide
* abstinence: if not sexually active, must commit to complete abstinence from intercourse

Female subjects, with the exception of those who are post-menopausal or surgically sterile, will undergo urine pregnancy tests approximately 7 days prior to first dose and approximately monthly.

* Diagnosis: An established clinical history of COPD in accordance with the definition of the American Thoracic Society (ATS).
* Severity of Disease: FEV1 post-albuterol/salbutamol at least 30 to no more than 80% of predicted normal and FEV1/FVC ratio post-albuterol/salbutamol of no more than 0.70 based on NHANES III reference values. Note that identical formulations of short-acting beta-agonist are called albuterol in the US and salbutamol in Canada.
* Smoking History: A history of smoking at least 10 pack-yr is required. Pack-yr are defined as the number of packs of cigarettes smoked per day multiplied by the number of yr smoked. Please note that both current and previous smokers are eligible for this study. Previous smoking is defined as no smoking for at least 6 months prior to consent; subjects are otherwise considered "current" smokers.
* CXR: Chest radiograph, within 1 yr prior to consent, without findings suspected to represent an active, clinically-significant process other than those believed to be related to uncomplicated COPD.
* Use of TIO: A history of using TIO with compliance at least 80% starting at least 14 days prior to V1, and ending 24 hr prior to V1, is required. Please note that any subject whose medical history precludes the safe use of TIO (such as significant narrow-angle glaucoma, known urinary retention, etc) should not be started on TIO for the purpose of this study.

Exclusion Criteria:

Subjects meeting any of the following criteria at V1 must not be enrolled in the study:

* Asthma: A current diagnosis of asthma.
* Other Diseases/Abnormalities: Any significant disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation, or which would affect the efficacy analysis if the disease/condition exacerbated during the study. Previously diagnosed cancer is considered a significant disease unless it is in complete remission for 2 yr (no evidence of tumor burden) at V1. Localized carcinomas of the skin that have been resected for cure are not exclusionary.
* Other Respiratory Disorders: Subject had lung resection surgery (e.g., lung volume reduction surgery or lobectomy) within 1 yr of V1 or has a significant respiratory disorder other than COPD (e.g., lung cancer, sarcoidosis, active tuberculosis, bronchiectasis, pulmonary fibrosis, sleep apnea, cystic fibrosis, or alpha-1-antitrypsin deficiency) that, in the opinion of the investigator, would put the safety of the subject at risk through study participation, or which would affect the efficacy analysis if the disease/condition exacerbated during the study.
* Acute Exacerbation of COPD: active disease within the past 6 wk. For the purpose of this study, an acute exacerbation of COPD will be identified using the following criteria [Anthonisen, 1987; Burge, 2003; Anzueto, 2009]: either
* worsening of two or more of the following "major" symptoms for at least two consecutive days:
* dyspnea
* sputum volume
* sputum purulence or
* worsening of any one major symptom together with any one of the following "minor" symptoms for at least two consecutive days:
* sore throat
* nasal discharge or nasal congestion
* fever without other cause
* increased cough or wheeze.
* Pulmonary Rehabilitation: Participation in the early, active phase of a Pulmonary Rehabilitation Program. For the purpose of this study, the "early, active" phase of pulmonary rehabilitation consists of sessions, scheduled on a regular and frequent basis (generally more than bi-weekly and for a total duration of at least 4 wk), held at an institution or at home, that include exercise training among interventions such as education and psychosocial support. Not included as the "early, active" phase of pulmonary rehabilitation are reinforcement or maintenance sessions that follow an "early, active" phase with interactions that are less frequent and less intense but may be scheduled for a longer total duration such as 6 months to 1 yr.
* 12-Lead ECG: Potential subjects are excluded if they have a functioning cardiac pacemaker. Otherwise, the investigator will determine the clinical significance of any ECG abnormality, and whether it precludes the potential subject from entering the study.
* Drug Allergy: Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, corticosteroid (intranasal, inhaled, or systemic including any components of the formulations [e.g. lactose or milk protein]), or atropine or its derivatives, including ipratropium or tiotropium.
* Body Mass Index (BMI): A BMI of 40 kg/m2 or higher.
* Use of ritonavir, ketoconazole or other potent inhibitors of CYP3A4: If any of these medications are used prior to V1, they must be stopped at V1 if indicated.
* Other Exclusionary medications: If any of the following medications are used prior to V1, they must be stopped as specified below.

(Medication, Washout period prior to V1) Any Investigational Drug, 30 days Oral or parenteral corticosteroids, 30 days ICS, 30 days ICS/LABA combination products (e.g., ADVAIR, Symbicort), 30 days Theophylline, 7 days Tiotropium, 24 hr LABA (e.g. formoterol or salmeterol), 12 hr Short-acting beta-agonists (e.g., albuterol or salbutamol), 6 hr Ipratropium or ipratropium-containing combination products (e.g., Combivent), 6 hr Oral beta-agonists, 6 hr

* Long-Term Oxygen Therapy (LTOT): Subject is on LTOT and is receiving supplemental oxygen more frequently than nocturnal-only.
* Affiliation with investigator site: Subject is a study Investigator, sub-Investigator, study coordinator, or employee of a participating Investigator or immediate family member of the aforementioned.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2010-07-19; Primary Completion 2011-05-01 (Actual); Study Completion 2011-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (27):
- United States (18):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Richmond, Virginia
- Canada (9):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Maltais F, Mahler DA, Pepin V, Nadreau E, Crater GD, Morris AN, Emmett AH, Ferro TJ. Effect of fluticasone propionate/salmeterol plus tiotropium versus tiotropium on walking endurance in COPD. Eur Respir J. 2013 Aug;42(2):539-41. doi: 10.1183/09031936.00074113. No abstract available. PMID 23904549
- [Derived] Borel B, Pepin V, Mahler DA, Nadreau E, Maltais F. Prospective validation of the endurance shuttle walking test in the context of bronchodilation in COPD. Eur Respir J. 2014 Nov;44(5):1166-76. doi: 10.1183/09031936.00024314. Epub 2014 Sep 3. PMID 25186261
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 113877 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113877 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113877 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113877 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113877 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113877 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113877 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the open-label 4-week run-in phase, participants received 18 micrograms Tiotropium (TIO) once daily. Participants completing this phase (n=255) were then randomized to receive either TIO+placebo or TIO+Fluticasone propionate/salmeterol combination DISKUS. The number enrolled in the protocol section reflects these 255 randomized participants.
Groups:
- Tiotropium (TIO): Tiotropium (TIO) was administered in the dose of 18 micrograms (mcg) once daily for a duration of 4 weeks
- TIO+Placebo: Matching placebo DISKUS twice daily (BD) plus tiotropium 18 mcg once daily for a duration of 4 weeks
- TIO+FSC: Fluticasone propionate/salmeterol combination (FSC) DISKUS, administered in the dose of 250/50 mcg BD, plus tiotropium in the dose of 18 mcg once daily for a duration of 4 weeks
Period: 4-Week Open-label Run-in Phase
Arm/Group | Tiotropium (TIO) | TIO+Placebo | TIO+FSC
Started | 338 | 0 | 0
Completed | 255 | 0 | 0
Not Completed | 83 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Did Not Meet Continuation Criteria | 61 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Period: 4-Week Double-blind Treatment Phase
Arm/Group | Tiotropium (TIO) | TIO+Placebo | TIO+FSC
Started | 0 | 131 | 124
Completed | 0 | 120 | 115
Not Completed | 0 | 11 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Adverse Event | 0 | 6 | 3
Not completed — Physician Decision | 0 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIO+Placebo | TIO+FSC | Total
Number analyzed (Participants) | 131 | 124 | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (9.85) | 62.5 (8.94) | 62.7 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 54 | 115
  Male | 70 | 70 | 140
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 4 | 10 | 14
  Japanese/East Asian Heritage/South East Asian | 1 | 2 | 3
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 126 | 110 | 236
  American Indian or Alaska Native and White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Exercise Endurance Time (EET) From Baseline (Week 3) to Week 8
Description: EET is defined as the time taken by a participant to exert himself during an exercise. EET was calculated based on the Endurance Shuttle Walk test (ESWT). The ESWT is a standardized, externally controlled, constant-paced field test for the assessment of endurance capacity in participants with chronic lung disease. Change from Baseline in EET was calculated as the value at Week 8 minus the value at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: Intent-to-Treat (ITT) Population: all participants randomized to study drug. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Seconds (sec)
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 122 | 115
Seconds (sec) | 23.3 (15.5) | 6.0 (16.2)
Statistical Analysis 1: Comparison: TIO+Placebo vs TIO+FSC; Test type: Superiority or Other; p = 0.181, ANCOVA — ANCOVA model with terms for treatment, investigator, Oxycon stratum, and baseline value; Mean Difference (Final Values) = -27.6, 95% CI 2-sided [-68.2 to 13.0], Standard Error of Mean 20.58

2. Secondary Outcome: Mean Change in Scores on the Exercise Dyspnea Scale (EDS) From Baseline (Week 3) to Week 8
Description: EDS is used to measure the level of breathlessness due to exercise, assessed using a 10-point modified Borg scale at 2-minute intervals during the ESWT: 0=no difficulty in breathing at all, 10=maximal breathing difficulty (BD). The participant pointed to the level on the scale correlating with his BD, and the local study coordinator confirmed that level verbally to him. Change from Baseline was calculated as the value at Week 8 minus the value at Baseline. A dyspnea score/time slope was calculated by fitting a linear regression line to the dyspnea scores reported during the exercise tests.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale/minute
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 121 | 110
Scores on a scale/minute | -0.1 (0.055) | -0.06 (0.058)

3. Secondary Outcome: Mean Change in EDS at Isotime From Baseline (Week 3) to Week 8
Description: EDS at isotime (last common time point for an exercise assessment [i.e., last Borg score time point of the shortest exercise test for each participant]) was assessed using a 10-point modified Borg scale. Change from Baseline in EDS at isotime was calculated as the value at Week 8 minus the value at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- TIO+Placebo: Matching placebo DISKUS BD plus tiotropium 18 mcg once daily for a duration of 4 weeks
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 121 | 110
Scores on a scale | -0.3 (0.2) | -0.5 (0.2)

4. Secondary Outcome: Mean Change in Pre-dose and Post-dose Resting Inspiratory Capacity (IC) From Baseline (Week 4) to Week 8
Description: Resting IC is the volume of gas that can be taken into the lungs in a full inhalation at the resting position. The resting IC was measured before and after dosing. Change from Baseline in pre-dose resting IC was calculated as the pre-dose value at Week 8 minus the pre-dose value at Week 4. Change from Baseline in post-dose resting IC was calculated as the post-dose value at Week 8 minus the pre-dose value at Week 4.
Time Frame: Baseline (Week 4) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Milliliters (mL)
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 122 | 115
Milliliters (mL)
  Pre-dose | -29 (29) | 60 (31.2)
  Post-dose | 73 (29.6) | 167 (31.4)

5. Secondary Outcome: Mean Change in Exercise Inspiratory Capacity (EIC) at the End of Exercise From Baseline (Week 3) to Week 8
Description: EIC is the volume of gas that can be taken into the lungs in a full inhalation during exercise. Participants were asked to undergo the IC test every 2 minutes during exercise and at the end of the exercise, to follow changes in operational lung volumes that occured in association with exercise. Change from Baseline in EIC was calculated as the value at the end of exercise at Week 8 minus the value at the end of exercise at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: mL
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 38 | 29
mL | -7.4 (120) | 46.6 (93.3)

6. Secondary Outcome: Mean Change in Flow of Oxygen (V'O2) Per Time Slope During the Course of the ESWT From Baseline (Week 3) to Week 8
Description: The V'O2 was measured during the ESWT using the Oxycon Mobile System (OMS), a portable telemetric monitoring system consisting of an oxygen sensor allowing for breath-by-breath measurement of gas exchange parameters in the lungs. The V'O2 was collected in units of mL and then regressed over the conduct of the exercise test measured in minutes. The V'O2 per time slope was calculated for each participant (par.) by fitting a linear regression line to the V'O2 recorded for each par. during the ESWT. V'O2 per time slope results were compared between treatment groups as means of these regression lin
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: mL/minute (min)
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 41 | 32
mL/minute (min) | -13.3 (10.36) | -6.1 (14.89)

7. Secondary Outcome: Mean Change in Flow of Carbon Dioxide (V'CO2) Per Time Slope During the Course of the ESWT From Baseline (Week 3) to Week 8
Description: The amount of CO2 in the hemoglobin of the participants was measured during the ESWT using the OMS. The system consisted of a carbon dioxide sensor and allowed breath-by-breath measurement of pulmonary gas exchange parameters. The V'CO2 per time slope was calculated for each participant by fitting a linear regression line to the V'CO2 recorded for each participant during the ESWT. V'CO2 per time slope results were compared between treatment groups as means of these regression lines. Change from Baseline in V'CO2 per time slope was calculated as the value at Week 8 minus the value at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 41 | 31
mL/min | -17.4 (10.36) | -0.7 (11.96)

8. Secondary Outcome: Mean Change in Minute Ventilation (V'E) Per Time Slope During the Course of the ESWT From Baseline (Week 3) to Week 8
Description: The V'E was measured in the participants during the ESWT using the OMS. The system consisted of a volume transducer, oxygen sensor, and carbon dioxide sensor and allowed breath-by-breath measurement of pulmonary gas exchange parameters. The V'E was collected in liters and then regressed over the conduct of the exercise test measured in minutes. The V'E per time slope was calculated for each participant by fitting a linear regression line to the V'E recorded for each participant during the ESWT. V'E per time slope results were compared between treatment groups as means of the regression lines.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liter (L)/min
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 42 | 34
Liter (L)/min | -0.7 (0.35) | -0.2 (0.49)

9. Secondary Outcome: Mean Change in Heart Rate (HR) Per Time Slope During the Course of the ESWT From Baseline (Week 3) to Week 8
Description: HR is defined as the number of heartbeats per unit of time, typically expressed as beats per minute (bpm). It was measured during the ESWT using the OMS. The HR was collected in units of bpm and then regressed over the conduct of the exercise test measured in minutes. The HR per time slope was calculated for each participant by fitting a linear regression line to the HR recorded for each participant during the exercise test. HR per time slope results were compared between treatment groups as means of these regression lines.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: bpm/min
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 42 | 34
bpm/min | -1.1 (0.70) | 0.7 (0.80)

10. Secondary Outcome: Mean Change in Respiratory Exchange Ratio (RER) Per Time Slope During the Course of the ESWT From Baseline to Week 8
Description: The respiratory exchange ratio was calculated as the ratio of VCO2 and VO2. The ratio of the amount of carbon dioxide and oxygen in the hemoglobin of the participants was measured during the ESWT using the OMS. The system consisted of oxygen and carbon dioxide sensors and allowed breath-by-breath measurement of pulmonary gas exchange parameters. Change from Baseline in RER was calculated as the value at Week 8 minus the value at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Ratio of VCO2 and VO2
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 42 | 34
Ratio of VCO2 and VO2 | -0.01 (0.004) | 0.01 (0.007)

11. Secondary Outcome: Mean Change in Respiratory Rate (RR) Per Time Slope During the Course of the ESWT From Baseline (Week 3) to Week 8
Description: RR is defined as the number of breaths taken within a set amount of time (typically within 60 secs). The RR of the participants was measured during the ESWT using the OMS. The system consisted of volume transducer oxygen and carbon dioxide sensors and allowed breath-by-breath measurement of pulmonary gas exchange parameters. The RR per time slope was calculated for each participant by fitting a linear regression line to the RR recorded for each participant during the ESWT. RR per time slope results were compared between treatment groups as means of these regression lines.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: breaths/min/min
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 42 | 34
breaths/min/min | -0.1 (0.18) | -0.5 (0.44)

12. Secondary Outcome: Mean Change in Respiratory Rate (RR) at Isotime During the Course of the ESWT From Baseline to Week 8
Description: RR is defined as the number of breaths taken within a set amount of time (typically within 60 secs). The RR of the participants at isotime was measured during the ESWT using the OMS. Change from Baseline in RR at isotime was calculated as the value at Week 8 minus the value at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: breaths/min
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 42 | 34
breaths/min | 0.8 (0.71) | -0.5 (0.68)

13. Secondary Outcome: Mean Change in Tidal Volume (VT) Per Time Slope During the Course of the ESWT From Baseline to Week 8
Description: VT is the lung volume representing the normal volume of air displaced between normal inspiration and expiration when extra effort is not applied (normal value is approximately 500 mL or 7 mL/kg body weight). VT was measured during the ESWT using the OMS, consisting of volume transducer O2 and CO2 sensors and allowing breath-by-breath measurement of pulmonary gas exchange parameters. The participant's VT per time slope was calculated by fitting a linear regression line (RL) to their VT during the ESWT. VT per time slope results were compared between treatment groups as means of these RLs.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: L/min
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 42 | 34
L/min | -0.02 (0.008) | 0 (0.014)

14. Secondary Outcome: Mean Change in Tidal Volume (VT) at Isotime During the Course of the ESWT From Baseline to Week 8
Description: VT is defined as the lung volume representing the normal volume of air displaced between normal inspiration and expiration when extra effort is not applied. The normal value is approximately 500 mL or 7 mL/kg body weight. The VT of the participants at isotime was measured during the ESWT using the OMS. Change from Baseline in VT at isotime was calculated as the value at Week 8 minus the value at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: L
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 42 | 34
L | -0.10 (0.04) | 0.08 (0.042)

15. Secondary Outcome: Mean Change in HR Per Time Slope During the Course of the ESWT Using Pulse Oximetry From Baseline to Week 8 (Non-OMS Subgroup)
Description: HR was measured during the course of the ESWT in the non-OMS subgroup using pulse oximetry. The HR per time slope was calculated for each participant by fitting a linear regression line to the HR recorded for each participant during the ESWT. HR per time slope results were compared between treatment groups as means of these regression lines. Change from Baseline in HR was calculated as the value at Week 8 minus the value at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed. A subgroup of participants specified sites provided cardio-respiratory and exercise IC measurements with the Oxycon Mobile System (OMS). Participants not at these sites formed the non-OMS subgroup.
Measure: Mean (Standard Error); unit: bpm/min
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 72 | 76
bpm/min | -0.8 (0.55) | -0.6 (0.56)

16. Secondary Outcome: Mean Change in Ratio of Respiratory Rate (RR) to Tidal Volume (VT) or RR/VT at Isotime During the Course of the ESWT From Baseline to Week 8
Description: The RR and VT of the participants at isotime were measured during the ESWT using the OMS. The ratio of RR per VT (value of RR divided by value of VT) at isotime was calculated. Change from Baseline in RR/VT at isotime was calculated as the value at Week 8 minus the value at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: breaths/min/L
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 42 | 34
breaths/min/L | 2.7 (1.14) | -2.5 (1.27)

17. Secondary Outcome: Mean Change in EIC at 2 to 3.5 Minutes During the Exercise Period From Baseline (Week 3) to Week 8
Description: The EIC was measured at 2 to 3.5 minutes during the exercise period. Change from Baseline in EIC was calculated as the value at Week 8 minus the value at Baseline.
Time Frame: Baseline (Week 3) and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: mL
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 24 | 22
mL | -148.3 (118.7) | 200 (110.2)

18. Secondary Outcome: Mean Change in Scores on the Chronic Respiratory Disease Questionnaire Self-Administered Standardized (CRQ-SAS) Questionnaire From Week 4 to Week 8
Description: The CRQ-SAS, a self-administered tool used to assess health-related quality-of-life (HRQOL), consists of 20 questions (q.) in 4 domains: Dyspnea (5 q.), Fatigue (4 q.), Emotional Function (7 q.), and Mastery (4 q.). Participants rated their experience on a 7-point scale in response to each q.: 1 (maximum impairment) to 7 (no impairment); higher scores indicate better HRQOL. Individual q. were equally weighted, and domain scores (range=1-7) were calculated as the mean across the non-missing items within each domain (domain scores were calculated although an individual item score was missing).
Time Frame: Week 4 and Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 122 | 115
Scores on a scale
  Mastery Score | 0.07 (0.08) | 0.09 (0.1)
  Fatigue Score | 0.11 (0.08) | 0.26 (0.1)
  Emotional Function Score | 0.10 (0.07) | 0.13 (0.08)
  Dyspnea Score | 0.21 (0.09) | 0.32 (0.1)

19. Secondary Outcome: Baseline Dyspnea Index (BDI) at Week 4 and Transition Dyspnea Index (TDI) at Week 8
Description: The BDI-TDI is a multidimensional dyspnea measurement. The BDI, administered at Week 4, consisted of 3 items (functional impairment, magnitude of task in exertional capacity, and magnitude of effort) requiring recall over the previous 4 weeks. BDI scores ranged from 0 (very severe impairment) to 4 (no impairment); the summed total score = 0 to 12. The TDI, administered at Week 8 as a follow-up of the BDI, consisted of the same 3 items requiring recall over the previous 4 weeks. TDI scores ranged from -3 (major deterioration) to +3 (major improvement); the summed total score = -9 to 9.
Time Frame: BDI: Week 4; TDI: Week 8
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | TIO+Placebo | TIO+FSC
Number analyzed (Participants) | 130 | 122
Scores on a scale
  BDI; n=130; 122 | 6.7 (0.20) | 6.9 (0.22)
  TDI; n=121, 115 | 1.1 (0.2) | 1.4 (0.2)

ADVERSE EVENTS:
Arm/Group | TIO+Placebo | TIO+FSC
Serious Adverse Events (participants affected / at risk) | 3/131 | 0/124
Other Adverse Events (participants affected / at risk) | 18/131 | 22/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIO+Placebo (N=131) | TIO+FSC (N=124)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIO+Placebo (N=131) | TIO+FSC (N=124)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dsyphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Chapped lips (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 0 | 2
Acute sinusitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.